CLINICAL TRIAL: NCT04751240
Title: Effect of Interval and Resistance Exercise on Physiological and Psychological Parameters.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Associate Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-323
Record Dates: First submitted 2021-02-07; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Body Composition
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: All subjects will participate in an exercise intervention consisting of sprint interval training and resistance training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIT and Resistance (Experimental): Participants will complete 10 weeks of a SIT and resistance training paradigm.
  Interventions: Behavioral: SIT and resistance training

INTERVENTIONS:
Behavioral: SIT and resistance training — Participants complete 30 sessions of sprints and resistance training. Outcomes are assessed acutely and at 6 months.

SUMMARY:
The purpose of this study is to examine the physiological and psychological effects of a sprint interval and resistance training intervention on females.

DETAILED DESCRIPTION:
Females aged 20-65 will attend 10 weeks of exercise training consisting of sprint interval training and resistance training for 30 sessions. We will examine changes in body composition, blood panel (fasting glucose, cholesterol, triglycerides), strength (bench press and back squat), aerobic capacity and psychological parameters (hardiness, affect, enjoyment, perception and self-regulation). The effects will be measured acutely after the program and 6-months after the cessation of the program.

ELIGIBILITY:
Inclusion Criteria:

* This population consists of: females, aged 25-55, who are: sedentary (not reporting a regular schedule of exercise over the last 3 months), and able to start an exercise program (assessed by the PARQ+)

Exclusion Criteria:

* Females who are below age 25 or over age 55, who are currently exercising and have existing conditions that would exclude them from exercise.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Fat mass post | Change in fat mass at 13 weeks
  Changes in Fat mass in Kg assessed by idexa
Fat mass retention | Change in fat mass at 6 months
  Changes in Fat mass in Kg assessed by idexa
Lean mass post | Change in lean mass at 13 weeks
  Changes in Lean mass in Kg assessed by idexa
Lean mass retention | Change in lean mass at 6 months
  Changes in Lean mass in Kg assessed by idexa
Visceral Fat post | Change in visceral fat at 13 weeks
  Changes in Visceral Fat in Kg assessed by idexa
Visceral Fat retention | Change in visceral fat at 13 weeks
  Changes in Visceral Fat in Kg assessed by idexa
Participate perception of the program post | 13 weeks
  Interviews to assess participants perception of the program
Participate perception of the program retention | 6 months
  Interviews to assess participants perception of the program

SECONDARY OUTCOMES:
Strength - bench press | Change in bench press at 13 weeks
  Changes in bench press measured in Kg
Strength - back squat | Change in back squat at 13 weeks
  Changes in back squat measured in Kg
Blood glucose post | Changes in fasting blood glucose at 13 weeks
  Changes in fasting blood glucose
Blood glucose retention | Changes in fasting blood glucose at 6 months
  Changes in fasting blood glucose
Cholesterol post | Changes in Cholesterol at 13 weeks
  Changes in Cholesterol
Cholesterol retention | Changes in Cholesterol at 6 months
  Changes in Cholesterol
Triglycerides post | Changes in Triglycerides at13 weeks
  Changes in Triglycerides
Triglycerides retention | Changes in Triglycerides at 6 months
  Changes in Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Wadsworth, PhD, Principal Investigator — Auburn University
Locations (1):
- School of Kinesiology, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shard with other researchers.